CLINICAL TRIAL: NCT06846814
Title: Second-Look Ultrasound Post Contrast-Enhanced Mammography for Additional Lesions Characterization
Status: Enrolling by invitation | Type: Observational
Sponsor: Graziella di Grezia (Other)
Collaborators: Link Campus University (Other); University of Campania Luigi Vanvitelli (Other)
Responsible Party: Sponsor-Investigator, Graziella di Grezia, Principal Investigator, Link Campus University
Organization: Link Campus University (Other)
Other Study IDs: T_4_2025
Record Dates: First submitted 2025-02-15; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer Diagnosis; Breast Cancer Detection
Keywords: Second look ultrasound; contrast enhanced mammography; breast cancer detection
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CEM protocol — The intervention consists of Second-Look Ultrasound (SLUS) performed following Contrast-Enhanced Mammography (CEM) to further evaluate additional lesions detected during routine breast imaging.
  When CEM identifies additional or suspicious lesions not clearly characterized by mammography alone, targeted ultrasound is conducted to assess lesion morphology, vascularity, and acoustic characteristics. Radiologists with expertise in both CEM and ultrasound interpretation will perform SLUS to determine whether the lesions require biopsy, short-term follow-up, or no further action. Findings will be correlated with histopathological results (if biopsy is performed) or follow-up imaging to assess diagnostic accuracy.

SUMMARY:
This study investigates the utility of second-look ultrasound (US) following contrast-enhanced mammography (CEM) to characterize additional lesions detected during routine breast imaging.

DETAILED DESCRIPTION:
The goal is to assess the diagnostic accuracy and clinical value of combining CEM with targeted ultrasound to improve lesion characterization and guide biopsy decisions.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients undergoing contrast-enhanced mammography for diagnostic or surveillance purposes.
* Identification of additional lesions on CEM requiring further evaluation.
* Ability to provide informed consent.

EXCLUSION CRITERIA:

* Known breast cancer diagnosis without suspicion of additional lesions.
* Contraindications to ultrasound or contrast agents.
* Patients with incomplete imaging data.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women aged 18 years and older undergoing CEM as part of diagnostic or surveillance protocols.
  Lesions detected by CEM that require additional characterization.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Detection Rate of Additional Lesions on CEM | Within 12 months of imaging assessment.
  This measure evaluates the number of additional lesions identified on Contrast-Enhanced Mammography (CEM) that require further assessment through second-look ultrasound or biopsy.

SECONDARY OUTCOMES:
Concordance Between Imaging Findings and Histopathology | Up to 3 months post-biopsy.
  This measure assesses the percentage of biopsied lesions in which imaging findings (from CEM and SLUS) correlate with the histopathological results
Concordance Between Imaging Findings and Follow-Up Imaging | 6-12 months after the initial CEM examination
  This measure evaluates the percentage of lesions that remain stable or resolve in follow-up imaging, confirming or refuting the initial CEM and ultrasound findings.

CONTACTS AND LOCATIONS:
Overall Officials: Graziella Di Grezia, Medicine, Principal Investigator — Link Campus University
Locations (1):
- University of Campania Luigi Vanvitelli, Naples, Italy

IPD SHARING:
Plan to Share IPD: No